CLINICAL TRIAL: NCT00515580
Title: Minimally Invasive Genioglossus And Hyoid Advancement For Obstructive Sleep Apnea Using Silhouette Sutures: A Pilot Study
Brief Title: Minimally Invasive Tongue Suture For Obstructive Sleep Apnea
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Results from first few subjects was not significantly improved over standard, traditional procedures.
Sponsor: West Side ENT (Other)
Responsible Party: Principal Investigator, Steven Y. Park M.D., Principal Investigator, West Side ENT
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NYEEI IRB 07.20
Record Dates: First submitted 2007-08-12; First posted 2007-08-14 (Estimated); Last update posted 2012-12-20 (Estimated); Status verified 2012-12

CONDITIONS: Obstructive Sleep Apnea; Upper Airway Resistance Syndrome
Keywords: obstructive sleep apnea; upper airway resistance syndrome; tongue suture; retrolingual tongue collapse; minimally invasive
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Mandibular Osteotomy; Suspensions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): Pilot study of 5 patients, with an additional 20 patients with conditional approval by the IRB once the initial 5 patient's data is reviewed.
  Interventions: Procedure: Tongue Sutures for Obstructive Sleep Apnea

INTERVENTIONS:
Procedure: Tongue Sutures for Obstructive Sleep Apnea — Mandibular osteotomy with placement of Silhouette sutures for genioglossus advancement and hyoid suspension.
  Other Names: tongue suture; mandibular osteotomy and genioglossus advancement; hyoid myotomy and suspension; uvulopalatopharyngoplasty (UPPP); obstructive sleep apnea

SUMMARY:
This is a pilot study to determine the usefulness of a newly developed, minimally invasive tongue suture procedure for people with obstructive sleep apnea.

DETAILED DESCRIPTION:
Obstructive sleep apnea is a common sleep-breathing disorder characterized by repetitive complete cessation of breathing due to pharyngeal obstruction. Untreated, it has been strongly associated with daytime sleepiness, hypertension, depression, coronary artery disease, stroke, and even death. It is estimated that up to 25% of men and 9% of women may suffer from this condition. One proposed mechanism of pharyngeal obstruction is that the posterior tongue is susceptible to collapse when supine during sleep, which causes further collapse of the soft palate and related structures. Treatment includes continuous positive airway pressure (CPAP), mandibular advancement devices, and various surgical options. There are many surgical options for treating tongue base collapse, many of which are morbid with significant pain and discomfort involved. Silhouette Sutures (Kolster Methods, Inc.) are designed to hold and grip soft tissues using intermittently placed dissolvable cones spaced by knots. It has been used widely for years for facial cosmetic procedures with excellent results and safety record. This is a pilot study evaluating the practicality and efficacy of using Silhouette Sutures in an innovative, minimally invasive technique that obviates the need for more aggressive and morbid procedures for obstructive sleep apnea.

ELIGIBILITY:
Inclusion Criteria:

Five patients will be recruited during a period of one year, or until a total of five patients have been recruited and have taken part. Patients must have undergone a formal overnight polysomnogram with documented obstructive sleep apnea within the past 2 years with no significant change in their weight or symptoms. They must have tried or refused all available nonsurgical options (CPAP or mandibular advancement devices), and must be ideal candidates for traditional upper airway surgery. Based on the polysomnogram results and specific entry criteria, patients will be recruited. All patients will undergo a full ENT examination and a fiberoptic laryngoscopy, examining the nasal cavity, palatal structures and tongue position, both in the sitting and supine positions (a routine part of the ENT examination).

Entry criteria include the following:

* men and women ages 18 to 65
* supine Park tongue position 3+ or greater
* tonsil size 2 or less
* Mueller's 2+ or less
* Friedman Stage II/III
* BMI ≤ 30
* AHI ≥ 5

Exclusion Criteria:

* Prior pharyngeal surgery
* History of radiation to the head and neck
* Dysmorphic facies or craniofacial syndrome
* ASA class IV or V
* Major depression or unstable psychiatric disorder
* Pregnancy
* Illiteracy (unable to complete required forms)
* No phone # or mailing address, or plans to change in 3 month period
* Any upper airway surgery within three month period

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2007-08; Primary Completion 2008-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Using standardized validated sleep disordered breathing and quality of life questionnaires (pre-op, 3 months, and 12 months). Patients will undergo a post-operative polysomnogram at 12 months. | one year or until 5 patients enrolled and completed

CONTACTS AND LOCATIONS:
Overall Officials: Steven Y. Park, MD, Principal Investigator — West Side ENT, PLLC
Locations (2):
- United States (2):
  - 330 West 58th Street, Suite 610, New York, New York
  - West Side ENT, New York, New York